CLINICAL TRIAL: NCT00263601
Title: A Multicentre, Placebo Controlled, Double-Blind Study for Evaluation of Safety and Efficacy of Preseasonal Specific Immunotherapy With an Allergoid Preparation of an Extract of a 6 Grass Pollen Mixture in Patients With Clinically Relevant Grass Pollen Sensitivity
Brief Title: Safety and Efficacy of Grass Pollen Allergoid in the Treatment of Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Al0101av
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Grass Pollen Allergy
Keywords: Allergovit; Grass pollen allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allergovit 6-grasses immunotherapy (Experimental): Seven injections (with 7 to 14 day intervals between each one) to reach maximum dose, followed by maintenance injections starting with 2 week intervals, followed by 4 week intervals until onset of the grass pollen season.
  Interventions: Biological: Allergovit 6-grasses
- Placebo (Placebo Comparator): Placebo injections was given the same way: Seven injections (with 7 to 14 day intervals between each one) to reach maximum dose, followed by maintenance injections starting with 2 week intervals, followed by 4 week intervals until onset of the grass pollen season.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Allergovit 6-grasses — Subcutaneous injections
  Other Names: Specific immunotherapy with an allergoid preparation.
  Arms: Allergovit 6-grasses immunotherapy
Other: Placebo — Subcutaneous injections
  Other Names: Comparator
  Arms: Placebo

SUMMARY:
The trial is performed to assess efficacy and safety of the Grass Pollen Allergoid in Allergic Rhinoconjunctivitis

DETAILED DESCRIPTION:
Pollen allergoids are prepared by chemical modification of partially purified native allergen aqueous extracts that have been depleted of components with a molecular mass of less than 5000 Daltons by diafiltration. Clinical studies have shown a good tolerance of aqueous grass, ragweed and tree pollen allergoids in comparison with allergen preparations. Adsorption of pollen allergoids onto aluminium hydroxide suspensions results in depot preparations which have been investigated in a series of clinical studies and shown to be well tolerated with good clinical efficacy. Depot pollen-allergoids were introduced into the German market in 1987 under the trade name Allergovit® and are now firmly established and recommended primarily for shortcourse preseasonal immunotherapy in pollinosis. Allergovit® is currently available in many European and non-European countries. A placebo-controlled study design was chosen as improvements in the symptoms of pollen allergies can not be shown over time, as pollen seasons of different years are not comparable. Due to the different mechanisms of action, specific immunotherapy can not be compared with anti-allergic drugs. Thus the only chance to prove efficacy for specific immunotherapy (SIT) is to test versus a parallel placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Positive Skin Prick test to grass pollen
* Positive RAST to grass pollen
* Positive specific provocation test to grass pollen

Exclusion Criteria:

* Serious chronic diseases
* Other perennial allergies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2001-11; Primary Completion 2004-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Symptom and Medication Score | Assessment after the first and second grass pollen season.
  The area under the curve (AUC) , derived from an analysis period of 42 days of the daily sum of the symptom and medication score (SMS).

SECONDARY OUTCOMES:
Rhinoconjunctivitis Quality-of-Life Questionnaire | First and second grass pollen season
  Changes in the scores of Rhinoconjunctivitis Quality-of-Life Questionnaire (RQLQ by E Juniper) at baseline (outside the grass pollen season), every two weeks during the 3 months grass pollen season (year 1+2).

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Narkus, M.D., Principal Investigator
Locations (1):
- Allergopharma GmbH & Co. KG, Reinbek, Germany

REFERENCES:
- [Result] Corrigan CJ, Kettner J, Doemer C, Cromwell O, Narkus A; Study Group. Efficacy and safety of preseasonal-specific immunotherapy with an aluminium-adsorbed six-grass pollen allergoid. Allergy. 2005 Jun;60(6):801-7. doi: 10.1111/j.1398-9995.2005.00790.x. PMID 15876311
- [Result] Williams A, Henzgen M, Rajakulasingam K. Additional benefit of a third year of specific grass pollen allergoid immunotherapy in patients with seasonal allergic rhinitis. Eur Ann Allergy Clin Immunol. 2007 Apr;39(4):123-6. PMID 17523386
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de